CLINICAL TRIAL: NCT00081133
Title: A Phase I/II Study to Determine Safety and Efficacy of Arsenic Trioxide (Trisneox™) in Combination With Imatinib (STI571, Gleevec™) in Patients With Chronic Myelogenous Leukemia in Accelerated or Blastic Phase Disease or Ph+ Acute Lymphoblastic Leukemia
Brief Title: Arsenic Trioxide and Imatinib Mesylate in Treating Patients With Accelerated Phase or Blastic Phase Chronic Myelogenous Leukemia or Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 03-126; CDR0000358923 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia
Keywords: accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Arsenic Trioxide; Imatinib Mesylate

INTERVENTIONS:
Drug: arsenic trioxide
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as arsenic trioxide, work in different ways to stop cancer cells from dividing so they stop growing or die. Imatinib mesylate may stop the growth of cancer cells by blocking the enzymes necessary for their growth. Combining arsenic trioxide with imatinib mesylate may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of arsenic trioxide when given with imatinib mesylate and to see how well they work in treating patients with accelerated phase or blastic phase chronic myelogenous leukemia or Philadelphia chromosome-positive acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolererated dose of arsenic trioxide when administered with imatinib mesylate in patients with accelerated or blastic phase chronic myelogenous leukemia or Philadelphia chromosome-positive acute lymphoblastic leukemia.
* Determine the rate of complete morphologic remission in the bone marrow of patients treated with this regimen.

OUTLINE: This is a phase I dose-escalation study of arsenic trioxide followed by a phase II study.

* Phase I:

  * Induction therapy: Patients receive oral imatinib mesylate once daily on days 1-35 (weeks 1-5) and arsenic trioxide IV over 1-4 hours on days 1-5, 8-12, 15-19, and 22-26 (weeks 1-4).

Patients undergo bone marrow evaluation on week 5. Patients achieving a morphologic remission proceed to consolidation therapy. Patients not achieving morphologic remission receive a second course of imatinib mesylate as above on weeks 6-10 and arsenic trioxide as above on weeks 6-9. Patients are re-evaluated on week 10. Patients achieving morphologic remission proceed to consolidation therapy. Patients not achieving a morphologic remission are removed from study.

* Consolidation therapy: Patients receive oral imatinib mesylate as in induction therapy on approximately weeks 6-11 (or weeks 11-16*) and arsenic trioxide IV over 1-4 hours on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26 (approximately weeks 6-9 OR weeks 11-14*).

Patients who remain in morphologic remission receive a second course of imatinib mesylate as in induction therapy on approximately weeks 12-17 (or weeks 17-22*) and arsenic trioxide as above (in consolidation therapy) on approximately weeks 12-15 (or weeks 17-20*).

NOTE: *For patients who receive a second course of induction therapy

Cohorts of 6 patients receive escalating doses of arsenic trioxide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive arsenic trioxide at the MTD and imatinib mesylate as in phase I.

Treatment in both phases continues in the absence of unacceptable toxicity or disease progression.

After completion of consolidation therapy, patients may continue imatinib mesylate off study at the discretion of the physician. Patients who become candidates for stem cell transplantation at any time during the study are removed from study.

PROJECTED ACCRUAL: A total of 6-43 patients (6-12 for phase I and 37 [including 6 patients from phase I] for phase II) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following:

  * Chronic myelogenous leukemia (CML) in one of the following phases:

    * Blastic phase*
    * Accelerated phase*

      * No appropriate donors for stem cell transplantation NOTE: *Must have received high-dose (600-800 mg/day) imatinib mesylate of no more than 3 months duration
  * Acute lymphoblastic leukemia

    * Philadelphia chromosome positive by cytogenetic confirmation

      * Patients with only bcr-abl-positive disease by polymerase chain reaction are not eligible
    * > 10% blasts in the bone marrow
* No isolated extramedullary disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN)
* AST ≤ 2 times ULN
* INR and PTT ≤ 1.5 times ULN (except for patients on anticoagulation therapy)

Renal

* Creatinine ≤ 2 times ULN

Cardiovascular

* Baseline QTc intervals < 480 ms
* No chronic arrhythmias
* No active coronary artery disease

Other

* No chronic electrolyte abnormalities
* No prior non-compliance to medical regimens
* No patients who are considered potentially unreliable
* No active serious infection
* No other active malignancies except superficial epithelial cancers
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for at least 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior peripheral blood stem cell or bone marrow transplantation

Chemotherapy

* Prior hydroxyurea allowed
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* More than 4 weeks since prior major surgery and recovered

Other

* Prior anagrelide allowed
* No concurrent warfarin for therapeutic anticoagulation

  * Concurrent low molecular weight heparin is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-12; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellin Berman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States